CLINICAL TRIAL: NCT06217471
Title: Role of Influenza A VIRus in the Biomolecular Pathogenesis of the Destabilization of Atherosclerotic Carotid Plaques
Brief Title: Influenza A VIRus and Destabilization of Atherosclerotic Carotid Plaques
Acronym: VIRAL
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Vascular Surgeon, Researcher, PI, IRCCS Policlinico S. Donato
Other Study IDs: VIRAL V1 - 131/int/2019
Record Dates: First submitted 2023-12-27; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — vascular atherosclerotic plaques, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Carotid Endoarterectomy — Surgical removal of atherosclerotic plaque from the carotid artery, collection of blood samples

SUMMARY:
Atherosclerosis is the main cause of cardiovascular diseases and is characterized by the accumulation of lipids and inflammatory cells such as macrophages and lymphocytes within the vessel wall of large and medium-sized arteries, forming so-called plaques. The underlying molecular mechanisms are not yet clearly understood. In particular, it is not yet clear what factors can cause the "destabilization" of atherosclerotic plaques, thus making them more vulnerable and prone to triggering acute cardiovascular events. Infectious agents have also been implicated in the pathogenesis of atherosclerosis. Some of them would be able to spread from the infected tissue and migrate to endothelial cells, promoting the secretion of inflammatory mediators and the oxidation of low-density lipoproteins (LDL), their accumulation in vascular cells and the formation of foam cells , fundamental mechanisms especially in the formation of vulnerable plaques.

Recently, many studies have shown that the influenza virus can also play a role in the destabilization of atherosclerotic plaques. However, the role of influenza A virus (IVA) infection and related vaccination in the destabilization of atherosclerotic plaques is still controversial. Furthermore, the underlying molecular mechanisms are still a matter of investigation.

Based on these data, we hypothesized that IV A infection may promote the destabilization of atherosclerotic plaques through a chronic postinfection immune response. This response would lead to systemic and local changes in the expression of pro-atherosclerotic cytokines and chemokines resulting in increased recruitment of monocyte macrophages and upregulation of the expression of scavenger receptors on the surface of macrophages with greater affinity for oxidized LDL (CD36 and Lectins- Like-oxLDL-receptor 1).

DETAILED DESCRIPTION:
The following data will be collected anonymously from the medical records:

* personal details (age, sex);
* comorbidity (presence of cardiovascular risk factors: arterial hypertension, smoking, dyslipidemia, ischemic heart disease, COPD, diabetes mellitus; chronic renal failure, history of cerebrovascular ischemic events);
* history of flu vaccination;
* clinical (weight, height); As per clinical practice, patients will undergo carotid endarterectomy surgery. Upon entry into the operating room, patients will be taken 4 ml of blood in 4 tubes with a specific anticoagulant (EDTA), from a peripheral venous access already positioned for the surgical procedure regardless of the study. These blood samples will be stored and processed appropriately for individual analyses.

Samples of atherosclerotic plaque removed during surgery will also be stored appropriately for subsequent investigations.

The data collected will be entered into the dedicated e-CRF and appropriately analyzed.

Use of blood samples Peripheral blood mononuclear cells (PBMC) will be separated and isolated from the venous blood sample using a Percoll gradient. These cells will be appropriately stimulated with influenza A virus antigens using specific commercial kits. This process will allow the evaluation of immune reactivity to the virus, both in the group of patients with vulnerable carotid plaque (group A) and in those with non-vulnerable plaque (group B). On the serum of the same samples, the quantitative expression of some cytokines/chemokines involved in inflammation and the atherosclerotic process (IL-6, IL-1β, TNF-α, IFN-γ, MCP-1) will be evaluated using the ELISA method).

The appropriate antibody evaluation will also be performed to test for any acute IV A infections.

Use of vascular samples Histology investigations will be carried out on atherosclerotic plaque samples which will allow determining the vulnerability or otherwise of the plaque, in such a way as to define the two groups of patients (A, vulnerable plaque; B, non-vulnerable plaque) to be analysed. and compare.

Western-Blot assays and immunohistochemical analyzes will also be performed on the same samples to evaluate the quantitative and qualitative expression of some molecules (V-CAM, I-CAM, E-Selectins) and receptors that identify scavenger macrophage cells (CD36 and Lectins -Like Ox-LDL-Receptor 1.

Finally, the same samples will be subjected to ELISA analysis for the quantitative research of the same cytokines/chemokines evaluated on the blood sample via RT-PCR. The possible presence of viral RNA will be evaluated on the atherosclerotic plaques by one step RT-PCR, as well as the T-specific cell reactivity to the IV A virus after the preparation of appropriate cell cultures which will be stimulated with the same commercial kit used to stimulate the PMBC of peripheral blood, according to the method described by Keller et al. Collaterally, the possible presence of viral or bacterial DNA in the plaques will be checked. In particular, the presence of DNA from Human Polyomaviruses and Human Herpesviruses (herpes simplex virus 7 and 2, varicella zoster virus, Epstein-Barr virus, human cytomegalovirus, human herpesvirus 6) and Chlamydia will be analyzed through Real Time PCR.

Evaluation of specific T-cell reactivity to virus IV A Taking as reference the method described by Keller et al, the stimulation index (SI) will be evaluated, both on the blood sample and on the atherosclerotic plaque, as the average count per minute (cpm) of cultures with the virus, divided by the mean cpm of parallel cultures without viruses.

Subsequently, the reactivity will be calculated based on the ratio between the SI of the plaque T cells and the SI of the peripheral blood T cells for each patient, defining responsive patients if the ratio is > 2 (patients with SI of the T cells T of the plaque significantly higher than those of the peripheral blood), and not responsive if the ratio is < 2 (in the latter case, patients with SI of the T cells of the peripheral blood greater than those of the plaque, or with SI of the T cells Plaque T not significantly higher than those of peripheral blood).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age > 18 years) who have given their consent to participate in the study, belonging to the Vascular Surgery Unit of the IRCCS Policlinico San Donato to undergo carotid endarterectomy surgery for significant carotid stenosis (in accordance with the Guidelines International guidelines, asymptomatic patients with carotid stenosis > 80% according to ECST and symptomatic patients with stenosis > 70% according to ECST

Exclusion Criteria:

* Minor patients
* Pregnant/breastfeeding women
* Patients who have not provided their consent to participate in the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients coming to the Vascular Surgery Unit of the IRCCS Policlinico San Donato to undergo carotid endarterectomy surgery for significant carotid stenosis
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
antigenic specificity of IV T cells | through study completion, an average of 3 years
  To test the antigenic specificity of IV T cells in carotid plaques and blood samples (peripheral blood mononuclear immune cells - PBMCs) of patients undergoing carotid endarterectomy (CEA) using the Stimulation Index, comparing results among a group of patients with vulnerable carotid plaque (group A) and a group of patients with stable plaque (group B, controls). Collaterally, the presence of viral RNA in the carotid plaques of patients in both groups will be evaluated; Blood samples will also be evaluated with serology for the presence of antibodies against IV A.
presence of viral RNA | through study completion, an average of 3 years
  The presence of viral RNA in the carotid plaques and in the blood of patients in both groups will be evaluated using real-time PCR.
expression of inflammatory chemokines/cytokines | through study completion, an average of 3 years
  Evaluate and compare the expression of inflammatory chemokines/cytokines involved in the recruitment and differentiation of monocytes (especially IL-6, IL-1β, TNF-α, IFN-γ, MCP-1), in the carotid plaque and in the blood peripheral of both groups; the results will be correlated to those obtained in objective 1.
expression of adhesion molecules and scavenger receptors | through study completion, an average of 3 years
  To evaluate and compare the expression of adhesion molecules and scavenger receptors with high affinity for oxLDL (CD36 and lectin-like oxLDL receptor) in carotid plaques between the two groups. The results will be correlated to those obtained in objectives 1 and 2.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Madjid M, Naghavi M, Litovsky S, Casscells SW. Influenza and cardiovascular disease: a new opportunity for prevention and the need for further studies. Circulation. 2003 Dec 2;108(22):2730-6. doi: 10.1161/01.CIR.0000102380.47012.92. Epub 2003 Nov 10. No abstract available. PMID 14610013
- [Result] Chistiakov DA, Melnichenko AA, Myasoedova VA, Grechko AV, Orekhov AN. Mechanisms of foam cell formation in atherosclerosis. J Mol Med (Berl). 2017 Nov;95(11):1153-1165. doi: 10.1007/s00109-017-1575-8. Epub 2017 Aug 7. PMID 28785870
- [Result] Guan X, Yang W, Sun X, Wang L, Ma B, Li H, Zhou J. Association of influenza virus infection and inflammatory cytokines with acute myocardial infarction. Inflamm Res. 2012 Jun;61(6):591-8. doi: 10.1007/s00011-012-0449-3. Epub 2012 Feb 29. PMID 22373653
- [Result] Keller TT, van der Meer JJ, Teeling P, van der Sluijs K, Idu MM, Rimmelzwaan GF, Levi M, van der Wal AC, de Boer OJ. Selective expansion of influenza A virus-specific T cells in symptomatic human carotid artery atherosclerotic plaques. Stroke. 2008 Jan;39(1):174-9. doi: 10.1161/STROKEAHA.107.491282. Epub 2007 Nov 29. PMID 18048854
- [Result] Haidari M, Wyde PR, Litovsky S, Vela D, Ali M, Casscells SW, Madjid M. Influenza virus directly infects, inflames, and resides in the arteries of atherosclerotic and normal mice. Atherosclerosis. 2010 Jan;208(1):90-6. doi: 10.1016/j.atherosclerosis.2009.07.028. Epub 2009 Jul 24. PMID 19665123
- [Result] Ricotta JJ, Aburahma A, Ascher E, Eskandari M, Faries P, Lal BK; Society for Vascular Surgery. Updated Society for Vascular Surgery guidelines for management of extracranial carotid disease. J Vasc Surg. 2011 Sep;54(3):e1-31. doi: 10.1016/j.jvs.2011.07.031. PMID 21889701